CLINICAL TRIAL: NCT04832139
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 4-PERIOD, 2-SEQUENCE, CROSSOVER STUDY TO EVALUATE THE BIOEQUIVALENCE OF MARSTACIMAB (PF-06741086) PREFILLED SYRINGE DEVICE AND PREFILLED PEN DEVICE FOLLOWING SUBCUTANEOUS ADMINISTRATION IN HEALTHY ADULT MALE PARTICIPANTS
Brief Title: A Study of Marstacimab to Compare Prefilled Pen (PFP) Device to Prefilled Syringe (PFS) Device
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in the benefit/risk assessment for the further administration of marstacimab in a healthy volunteer population.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7841009; 2020-004369-38 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; Phase 1; Prefilled Pen; Prefilled syringe; pharmacokinetic; subcutaneous; hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Marstacimab Prefilled Pen (PFP), then marstacimab Preflled Syringe (PFS) (Experimental): Participants will first receive single dose PFP, then PFS, then repeating single dose PFP, then single dose PFS with a minimum of 21 days between single doses.
  Interventions: Drug: Marstacimab PFP; Drug: Marstacimab PFS
- Marstacimab PFS, then marstacimab PFP (Experimental): Participants will first receive single dose PFS, then PFP, then repeating single dose PFS, then single dose PFP with a minimum of 21 days between single doses.
  Interventions: Drug: Marstacimab PFP; Drug: Marstacimab PFS

INTERVENTIONS:
Drug: Marstacimab PFP — 300 milligrams (mg) subcutaneous injection marstacimab PFP
  Other Names: PF-06741086
Drug: Marstacimab PFS — 300 mg subcutaneous injection of marstacimab PFS
  Other Names: PF-06741086

SUMMARY:
The goal in this study is to show that there are not significant differences in biologic activity of the study drug when administered using either the prefilled pen and prefilled syringe.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight ≥ 50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease
* Any condition possibly affecting drug absorption (eg, conditions affecting SC administration)
* Previous or current treatment for and/or history of coronary artery diseases, venous or arterial thrombosis, or ischemic disease.
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb or HCVAb
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior, laboratory abnormality or COVID-19 related condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test at screening and/or admission
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic)
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening:

  * AST or ALT level ≥1.5 × ULN;
  * Total bilirubin level ≥1.5 × ULN.
* An estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m2 based on the CKD-EPI equation.
* Resistance to activated protein C (or Factor V Leiden mutation), prothrombin 20210 mutation, antithrombin III deficiency, protein C deficiency, or protein S deficiency.
* Presence of Lupus anticoagulant anti-cardiolipin antibodies (IgG, IgM or IgA)
* High sensitivity C-reactive protein (hsCRP) above the upper limits of normal
* Abnormal hematology values as defined by the following laboratory tests at Screening and/or admission:

  * Platelet count <100,000/uL
  * Hemoglobin level <10 g/dL
* A positive COVID-19 test.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening
* Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of the protocol
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Area Under the plasma concentraiton time Curve from time zero extrapolated to infinite time (AUCinf) | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Maximum observed plasma concentration (Cmax) | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose

SECONDARY OUTCOMES:
Area under the concentration time curve from time 0 to time of last quatifiable concenteration | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Time for Cmax | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Apparent clearance after subcutaneous dose | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Apparent volume of distribution after subcutaneous dose | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Terminal half-life after subcutaneous dose | Day 1 Hour 0, 1, 2, 4, 8, 12, 24, 48, 72; Day 7; Day 14; Day 21 after each dose
Incidence of clinically significant laboratory value abnormalities | Baseline through the end of study, approximately 161 days
Incidence of anti-drug antibody against marstacimab | From Day 1, Period 1 through Day 21, Period 4 over a total of 84 days
Incidence of Adverse Events | Baseline through the end of study, approximately 161 days
Incidence of neutralizing antibody against marstacimab | From Day 1, Period 1 through Day 21, Period 4 over a total of 84 days
Incidence of Serious Adverse Events | Baseline through the end of study, approximately 161 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841009